CLINICAL TRIAL: NCT04922827
Title: A Randomized, Controlled, Multicenter, Open Label Phase II Clinical Study to Evaluate Infliximab in the Treatment of Patients With Severe COVID-19 Disease
Brief Title: Infliximab in the Treatment of Patients With Severe COVID-19 Disease
Acronym: INFLIXCOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZKSJ0137_INFLIXCOVID; 2021-002098-25 (EudraCT Number)
Record Dates: First submitted 2021-06-10; First posted 2021-06-11 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Infliximab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infliximab + Standard of Care (Experimental)
  Interventions: Drug: Infliximab; Other: Standard of Care
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Infliximab — single intravenous administration of 5 milligrams/kilogram
  Arms: Infliximab + Standard of Care
Other: Standard of Care — Standard of Care

SUMMARY:
In this trial, patients that are severely affected by the disease COVID-19 will either receive infliximab, an anti-inflammatory drug, or standard therapy. Infliximab is a drug that inhibits inflammation by blocking a molecule called TNFα. The patients receive the drug via an infusion into a vein. The primary goal of this trial is to see whether the drug infliximab affects how many people died from COVID-19 after 28 days by comparing patients receiving the drug in addition to standard therapy with patients only receiving standard therapy.

Furthermore, this trial will look at whether the drug is safe to use in these patients, whether it has an effect on the inflammation and whether it can affect how ill patients are after surviving the disease.

The trial is conducted in more than one hospital. As COVID-19 is responsible for a global pandemic, positive results of this trial could affect patients, healthcare and economic systems worldwide.

DETAILED DESCRIPTION:
The long-term goal of this research project is to develop a new pharmacological treatment strategy for patients with COVID-19. Its primary aim is the assessment of efficacy and safety of the TNFα antibody infliximab in the treatment of patients with severe COVID-19 in a phase-2 trial. Infliximab is expected to attenuate the inflammatory reaction in patients and thereby positively influence the course of the disease.

The primary endpoint is the difference in 28-day-mortality of patients with severe COVID-19 receiving one dose of 5mg per kg body weight infliximab intravenously in addition to the standard of care (intervention group) compared with patients receiving standard of care (control group).

Secondary aims of this trial include the assessment of the safety of the TNFα antibody infliximab in the treatment of patients with severe COVID-19, of its effect on an excessive immune response and of its effect on the morbidity and prognosis as well as the characterization of the analytical cohorts.

The multi-centre design facilitates the transferability of study results to hospitals of similar healthcare level. Should infliximab prove to be superior to standard therapy, this could be reflected in a reduced disease severity and mortality.

The results of this study could influence the therapy of patients with COVID-19 worldwide and affect the course of the disease worldwide, as infliximab is approved by several international drug agencies and globally available. Due to the high incidence of COVID-19 worldwide and the immense effects of the pandemic on societies, health care and economic systems, any progress in the treatment of this new disease would constitute a great success. This would not only impact individual patients but also have positive economic effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Infection with SARS-CoV-2 (virus detection by means of a PCR test not older than 72 hours)
* Bipulmonary infiltrates (detection by means of X-rays or computed tomography)
* COVID inflammation score ≥ 10
* Ferritin concentration (serum or plasma) ≥ 500 ng / ml
* Arterial oxygen saturation ≤ 93% when breathing room air
* written informed consent from the patient
* Potentially childbearing women: negative pregnancy test

Exclusion Criteria (in medical history):

Contraindications study medication:

* Hypersensitivity to the active substance infliximab (or any of the other ingredients of the medicine) or to other murine proteins
* active or latent tuberculosis
* acute or chronic hepatitis B
* severe infections such as invasive fungal infections, bacterial sepsis, or abscesses
* opportunistic infections (e.g. pneumocystosis, listeriosis)
* moderate or severe heart failure (NYHA class III / IV)
* Immunosuppression (e.g. organ transplantation, AIDS, leukopenia)
* Malignancies or lymphoproliferative diseases or chemotherapy within the last 4 weeks
* Multiple sclerosis or peripheral demyelinating diseases, including the Guillain-Barré syndrome
* Treatment with other biologics for therapy for approved indications of infliximab (e.g. for rheumatoid arthritis, Crohn's disease, ulcerative colitis, ankylosing spondylitis, psoriatic arthritis, psoriasis)

Further exclusion criteria:

* Autoimmune disease with biologics therapy
* Current treatment with TNF antibodies, convalescent plasma, bamlanivimab, or other experimental treatments for COVID-19
* High-flow oxygen therapy, non-invasive / invasive ventilation (WHO-COVID-19 PROGRESSION Scale > 5)
* pre-existing long-term ventilation or home oxygen therapy
* Child-Pugh C liver cirrhosis
* Pregnancy or breastfeeding
* Patients with a life expectancy < 90 days due to other medical conditions
* Limitation or discontinuation of therapy (e.g. refusal of artificial ventilation)
* Participation in another interventional study
* Previous participation in this study
* Interdependence between the patient and the coordinating investigator or other members of the study team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28 days after randomization
  differences in mortality-rates between both study arms (Infliximab + Standard of Care vs. Standard of Care) 28 days after randomisation

SECONDARY OUTCOMES:
safety of Infliximab administration | up to 90 days after randomization
  frequencies of adverse events (AEs) and serious adverse events (SAEs)
assessment of the effect of infliximab on an excessive immune response in patients with COVID-19: Interleukin 6 | day 7 and day 14 after randomization
  change in the interleukin-6 (IL-6) concentration in the blood from randomization to day 7 and day 14 after randomization
assessment of the effect of infliximab on an excessive immune response in patients with COVID-19: ferritin | day 7 and day 14 after randomization
  change in the ferritin concentration in the blood from randomization to day 7 and day 14 after randomization
assessment of the effect of infliximab on an excessive immune response in patients with COVID-19: lymphocyte count | day 7 and day 14 after randomization
  change in the lymphocyte count from randomization to day 7 and day 14 after randomization
assessment of the severity and frequency of organ failure: ventilation-free days | day 28 after randomization
  ventilation-free days until 28 days after randomization
assessment of the severity and frequency of organ failure: renal replacement therapy-free days | day 28 after randomization
  renal replacement therapy-free days until 28 days after randomization
assessment of the severity and frequency of organ failure: vasopressor-free days | day 28 after randomization
  vasopressor-free days until 28 days after randomization
occurence of Acute Respiratory Distress Syndrome (ARDS) | day 28 after randomization
  rate of occurrence of ARDS until 28 days after randomization
WHO-COVID-19-Progression Scale | day 7, 14 and 28 after randomization
  WHO-COVID-19-Progression Scale on day 7, 14 and 28 after randomization
rate of admission to the intensive care unit | day 28 after randomization
  rate of admission to the intensive care unit after randomization up to day 28
length of stay: hospital | day 28 after randomization
  length of hospital stay up to day 28 after randomization
length of stay: intensive care unit | day 28 after randomization
  length of intensive care unit stay up to day 28 after randomization
mortality | day 14 and 90 after randomization
  mortality rates 14 and 90 days after randomization
health related quality of life: visual analogue scale | day 90 after randomization
  EQ5D-3L: visual analog scale value 90 days after randomization
health related quality of life: index | day 90 after randomization
  EQ5D-3L: index value 90 days after randomization
incidence of cardiomyopathy | day 3 and 7 after randomization
  incidence of cardiomyopathy 3 and/or 7 days after randomization

OTHER OUTCOMES:
collection and storage of blood and urine sample | day 3, 7 and 14 after randomization
  collection and storage of blood and urine sample for the investigation of translational research questions by analysing biomarkers of organ, metabolic and immunological function and regulation
comparison with other cohorts | up to day 90 after randomization
  comparison of the course of disease of patients with severe COVID-19 and previously generated datasets from patients with sepsis and health subjects

CONTACTS AND LOCATIONS:
Overall Officials: Sina M Coldewey, Prof. Dr. Dr. med., Principal Investigator — Department of Anaesthesiology and Intensive Care Medicine, Jena University Hospital; Andreas Stallmach, Prof. Dr. med., Principal Investigator — Department of Internal Medicine IV (Gastroenterology, Hepatology, and Infectious Diseases), Jena University Hospital
Locations (4):
- Germany (4):
  - Universitätsklinikum Knappschaftskrankenhaus Bochum, Bochum
  - Klinikum Fulda, Fulda
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Jena University Hospital, Jena

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coldewey SM, Neu C, Bloos F, Baumbach P, Schumacher U, Bauer M, Reuken P, Stallmach A. Infliximab in the treatment of patients with severe COVID-19 (INFLIXCOVID): protocol for a randomised, controlled, multicentre, open-label phase II clinical study. Trials. 2022 Sep 2;23(1):737. doi: 10.1186/s13063-022-06566-5. PMID 36056419